CLINICAL TRIAL: NCT03308903
Title: Can the Sit-to-Stand Test be Used as a Screening Tool to Detect Sarcopenia in Community-dwelling Older People?
Brief Title: Use of the Sit-To-Stand Task as a Screening Tool for Sarcopenia The
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Prof David Hewson, Professor of Health and Ageing, University of Bedfordshire
Other Study IDs: IHREC751
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: DEXA scan — The participant will undergo a whole-body DEXA (DEXA; GE Medical Systems, Chalfont St Giles, UK) scan, lasting approximately 5 minutes. This scan will produce body composition data, including estimates of lean body mass (LBM), appendicular lean mass (aLM) and body fat percentage (BF%).

SUMMARY:
A common condition associated with ageing is sarcopenia, which is a progressive decrease in muscle mass. Sarcopenia is associated with adverse outcomes including increased mortality, and places a major burden on healthcare spending, with the annual cost of sarcopenia in the United States exceeding that of osteoporosis and hip fracture. In the UK, the prevalence of sarcopenia in community-dwelling older people has been estimated at 5% for men and 8% for women. Current guidelines for sarcopenia diagnosis require muscle mass to be measured using costly devices such as Dual Energy X-ray Absorptiometry (DXA) and Magnetic Resonance Imaging (MRI). Previous research has found strong relationships between the sit-to-stand (STS) test and both muscle mass and muscle strength. This pilot study aims to examine this relationship in community-dwelling older people to develop predictive equations for initial screening of sarcopenia.

Forty subjects will be tested using the diagnostic criteria developed by the European Working Group on Sarcopenia in Older People (EWGSOP). Muscle mass will be measured using the DXA and diagnostic ultrasound. Muscle strength will be measured using isokinetic dynamometer, handgrip dynamometry, and hand-held dynamometry. Functional performance will be measured using the Timed-up-and-Go and gait velocity, and the STS. Subjects will perform two variants of the STS; the five times STS (5STS), which requires subjects to perform five consecutive STS movements as quick as possible, and the 30-second STS (30STS), which requires subjects to perform as many STS movements as possible in 30 seconds. All testing will be completed in a single session lasting 90 minutes for each subject. Testing will be performed at the University of Bedfordshire Polhill Campus. Subject recruitment will be recruited using advertisement posters and word of mouth.

DETAILED DESCRIPTION:
Loss of function and mobility becomes an increasing concern as we age. Life expectancy is continuing to increase, which in turn leads to age-related diseases and syndromes becoming more common, complex and costly. Sarcopenia is the deficiency of muscle and this refers to the gradual loss of skeletal muscle mass and strength that occurs with advancing age This age-related disease is now understood as a major clinical problem for the elderly and it is becoming a public health issue in today's society.

The European Working Group on Sarcopenia in Older People (EWGSOP) has developed a clinical and practical definition and a diagnostic criterion for age-related sarcopenia. They define sarcopenia as "a syndrome characterised by progressive and generalised loss of skeletal muscle mass and strength with a risk of adverse outcomes". The EWGSOP further develop their definition of sarcopenia into two different categories and three different stages. The two categories are known as primary sarcopenia and secondary sarcopenia. Primary or age-related sarcopenia is when there is no other cause evident except ageing. Whereas secondary sarcopenia is when there are one or more other causes, such as activity-related, disease-related or nutrition-related. The three stages of sarcopenia reflect the severity of the condition; these are known as presarcopenia, sarcopenia and severe sarcopenia. The presarcopenia stage is described as having low muscle mass, without influencing muscle strength or physical performance. The sarcopenia stage is indicated by again having low muscle mass plus either having low muscle strength or poor physical performance. The severe sarcopenia stage is characterised by meeting all three criteria of the definition; low muscle mass, low muscle strength and poor physical performance. The EWGSOP specify that the measurable variables of sarcopenia are muscle mass, muscle strength and physical performance. The challenge they raised is the difficulty determining which methods are best to accurately measure these variables.

The EWGSOP indicate that muscle mass is best measured using body imaging techniques such as magnetic resonance imaging (MRI) or computer-tomography (CT). Both MRI and CT scans are known as the gold standards for measuring muscle mass within research. However, they are costly procedures that are not always freely available. Muscle mass can also be measured through dual energy X-ray absorptiometry (DEXA), for determining the presence of and formulating a diagnosis of sarcopenia. DEXA is based on the measurement of X-ray transmission crossing human tissues. The radiation energies produced by the DEXA are variably attenuated, either scattered or absorbed, by the anatomical structures within the body, dependent on the intensity of the energy and the density and thickness of the human tissues. DEXA enables measurements of fat mass (FM), lean mass (LM) and bone mineral content (BMC) and can assess body masses and bone mineral density (BMD) on a regional and a whole-body basis, whilst exposing only minimal radiation to the patient. According to the EWGSOP, DEXA is a preferred alternative method for measuring muscle mass within research and clinical use. However, it has been reported that measures of muscle mass from DEXA scans do not seem to be accurate, with a site-specific assessment of loss of muscle mass, using ultrasound-based assessment suggested. Ultrasound has been reported to be an effective and non-invasive tool to determine muscle wasting, potentially leading to an earlier and more accurate detection of sarcopenia.

Measures of muscle mass are not as good a predictor of physical capability as muscle strength. Lower limb muscle strength is more relevant for gait and physical function than upper limb muscle strength. However, the EWGSOP recognise handgrip strength as the most widely used method for measuring muscle strength to screen for sarcopenia. Handgrip strength is strongly related with lower extremity muscle power, knee extension torque and calf cross-sectional muscle area. Consequently, it has been documented that muscle power deteriorates earlier and quicker than muscle strength in older populations. Therefore, a measure of muscle power could be more beneficial in the diagnosis of sarcopenia as older people lose power quicker than they do strength. Isokinetic dynamometers (IKD) are a commonly used tool and are recognised as a gold standard measure of muscle power and strength. IKD's measure force dynamically through a specified range of motion whilst allowing the velocity of the movement to be controlled and measured. It is recognised as a popular method to assess muscle function in both clinical and research settings. However, due to IKD's not being portable and are not always accessible, there has been a rise in the use of hand-held dynamometry (HHD) to assess isometric muscle strength. It has been reported that HHD is a simple and inexpensive and a reliable and valid assessment tool for measuring strength, particularity in older adults. The use of isometric strength testing may be more suitable for older adults if there is a limited range of joint motion and if joint pain is prevalent, concentric actions may be challenging.

The importance of using physical performance measures within clinical geriatrics as well as ageing research has also been documented. There are many tests of physical performance that have been validated and are widely used. The EWGSOP identified popular methods for evaluating physical performance. These include the Short Physical Performance Battery (SPPB), usual gait speed (GS), the timed get-up-and-go (TUG) test and the stair climb power test. The ability to rise from a chair has been used in clinical evaluations and on-going assessments for decades. This everyday task was standardised and developed into the 'timed-stands' test. This test was initially designed to measure functional strength of the lower extremities as participants completed 10 timed-stands. Variations of this sit-to-stand (STS) task have evolved and now one of the most commonly used tools for clinical evaluation of physical performance is the Five-Times-Sit-To-Stand (5STS) test. The 5STS, requires the participant to stand up and sit down from a chair five times, with performance taken as the time to complete the test. The STS task was modified further, with a standardised 'time' protocol of 30 seconds (30sSTS), requiring the participant to stand up and sit down as many times as possible within 30 seconds. They reasoned the use of the 30sSTS instead of participants performing a predetermined number of repetitions (e.g. 5STS, 10STS) to assess a wider range of ability. Moreover, the 5STS and potentially even the 10STS can be recorded as the participant performs the 30sSTS. In addition to functional performance, the STS task could also be used to estimate muscle power and even muscle mass. In a recent study, an accurate estimation of lower-limb muscle power was obtained using a simple regression equation in which only body weight and the number of STS performed in 20 seconds, of a 30-second trial were used. Another study had also reported a good estimation of muscle mass obtained from an MRI, again using a simple regression equation in which only three basic variables were used, namely leg length, body mass and the time taken for a single STS movement.

Research Aim The aim of this study is to validate the use of the Sit-To-Stand task as a measure of muscle mass, muscle strength and power and physical performance in screening for sarcopenia compared to gold standard measures, in older adults aged 65 years and over.

Research Objectives

1. Suitability of the Sit-To-Stand task as a measure of muscle mass in comparison to the gold standard equivalents, the dual energy x-ray absorptiometry scan and diagnostic ultrasound.
2. Suitability of the Sit-To-Stand task as a measure of muscle strength and power in comparison to the gold standard equivalents, the isokinetic dynamometer the hand-grip strength dynamometer and the hand-held dynamometer.
3. Suitability of the Sit-To-Stand task as a measure of physical performance in comparison to other well used physical function tests, the Timed-Up-and-Go and gait.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Community-dwelling adults
* Aged 65+ years

Exclusion Criteria:

* Cardiovascular and/or respiratory problems
* High blood pressure (140/90mmHG or higher)
* Low blood pressure (90/60mmHg or lower)
* A diagnosis of arthritis and/or osteoporosis
* Had a musculoskeletal injury within the last twelve months
* Had an X-ray examination with contrast medium in the 3 weeks prior to the DEXA scan (if this does apply to the participant, the date of which they will participate will be delayed until 3 weeks after the date of their contrast scan)
* Recently had a Nuclear Medicine diagnostic or therapy investigation, depending on its nature (this will be referred to the Medical Physics Expert to determine if and when the participant can receive a DEXA scan for this study)
* Any significant internal metalwork or irremovable external metalwork.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling people aged 65 years and over with no musculoskeletal problems.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mass measurement using dual X-ray absorptiometry | 5 minutes
  The participant will undergo a whole-body DEXA (DEXA; GE Medical Systems, Chalfont St Giles, UK) scan, lasting approximately 5 minutes. This scan will produce body composition data, including M and body fat percentage (BF%). For the purpose of this study, aLM values will be calculated in relation to height (sum of LBM in the arms and legs, scaled to height) (aLM/ht²).

SECONDARY OUTCOMES:
Hip and knee flexion and extension and ankle plantarflexion and dorsiflexion of both lower extremities on the Biodex System 3 Isokinetic Dynamometer | 5 minutes
  Participants will perform two sets of five repetitions of hip and knee flexion and extension and ankle plantarflexion and dorsiflexion of both lower extremities on the Biodex System 3 Isokinetic Dynamometer (IKD) (Suffolk, UK), with a 2-minute rest period between sets. The angular velocity of the IKD will be set at 60º/s.
Five times sit to stand test | 5 minutes
  Participants will sit in a straight back chair with a solid seat that is 16" high. Participants will have their arms folded across their chest. They will then stand up and sit down as quickly as possible five times, keeping their arms folded across their chest. The test is measured with a stopwatch and is completed when the participant stands for the 5th time.
Diagnostic ultrasound | 5 minutes
  Sonographic estimates of LBM will be measured using a diagnostic ultrasound. Muscle thickness measurements will be taken from both arms and legs of the participants.
Grip strength | 5 minutes
  A measure of handgrip strength will be taken using the JAMAR PLUS + (Patterson Medical, IL, USA) of both the participant's upper extremities. Measures will be taken twice with a 2-minute rest period between trials. This requires the participant to exert their maximal grip in an isometric contraction.
Handheld dynamometer assessment of muscle strength | 5 minutes
  Measures of isometric muscle strength will be measured using the hand-held dynamometer (HHD). Measures will be taken from the hip flexors, quadriceps, hamstrings, gastroc-soleus complex and tibialis anterior of both lower extremities.
Timed Up and Go test | 2 minutes
  The participant sits on a standard armchair, placing his/her back against the chair and resting his/her arms chair's arms. The participant is instructed to use a comfortable and safe walking speed. The participant walks to a line that is 3 meters away, turns around at the line, walks back to the chair, and sits down. The test ends when the patient's buttocks touch the seat.
  A stopwatch is used to time the test (in seconds).
30-second sit to stand test | 5 minutes
  Participants will sit in a straight back chair with a solid seat that is 16" high. Participants will have their arms folded across their chest. They will then stand up and sit down as quickly as possible for 30 seconds, keeping their arms folded across their chest. The test is measured with a stopwatch and is completed after 30 seconds, with the number of completed sit to stands taken as the score.
Gait velocity | 2 minutes
  Participants will be asked to walk at a comfortable pace between two lines, marked five metres apart. The time taken will be measured with a stopwatch, with total time taken as the score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bedfordshire, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided